CLINICAL TRIAL: NCT04440332
Title: The Clinical Significance of Surveillance of Lymphocyte and Immunocyte Subsets in Peripheral Blood of Esophageal Squamous Cell Carcinoma Patients With Neoadjuvant Chemoradiotherapy Combine Surgery or Surgery Alone (pLINE）.
Brief Title: Surveillance of Peripheral Blood of Lymphocyte and Immunocyte in Neoadjuvant Therapy Patients With Esophageal Squamous Cell Carcinoma (pLINE)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Yongtao Han, Director,Head of Thoracic Surgery, Sichuan Cancer Hospital and Research Institute
Other Study IDs: 3001
Record Dates: First submitted 2020-06-08; First posted 2020-06-19 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Esophageal Squamous Cell Carcinoma; Neoadjuvant Therapy; Surgery
Keywords: esophageal squamous cell carcinoma; lymphocyte subsets; neoadjuvant chemoradiotherapy; immunocyte
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Neoadjuvant chemoradiotherapy treatment represents the standard approach for resectable locally advanced esophageal squamous cell carcinoma. The incidence of pulmonary infection and other perioperative complications were higher in patients who received esophagectomy and neoadjuvant chemoradiotherapy than those without neoadjuvant treatment and surgery patients. However, reliable clinical data can quantify the damage degree of immunologic function caused by chemotherapy and radiotherapy is still unknown. This project regards the level of lymphocyte and immunocyte in peripheral blood as a quantitative index to reflect the dynamic change of the immunologic function of patients with locally advanced esophageal squamous cell carcinoma after neoadjuvant chemoradiotherapy treatment. Meanwhile, the investigators will also investigate the relationship between the level of lymphocyte and immunocyte in peripheral blood and the response rate of neoadjuvant therapy.

DETAILED DESCRIPTION:
Peripheral blood will be collected from patients who will undergo esophagectomy and/or neoadjuvant therapy. The setting time is before chemoradiotherapy, finishing chemoradiotherapy, pre-operation, postoperative day 1, day 3, day 5, and day 7. These blood samples will be used for detection and analysis in lymphocyte and immunocyte by flow cytometry.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histologically confirmed locally advanced resectable thoracic ESCC; and requires esophagectomy alone or neoadjuvant chemoradiotherapy combined surgery treatment; Clinical stage T1-3N2-3M0 (AJCC 8 TNM classification);
* 2. At least one measurable lesion in accordance with RECIST 1.1;
* 3. Have a performance status of 0 or 1 on the ECOG Performance Scale;
* 4. Expected survival time is greater than 6 months;
* 5. Good organ function level: Hematology: white blood cell ≥3×10^9/L, neutrophil ≥1.5×10^9/L, hemoglobin ≥90 g/L and platelet ≥100×10^9/L; hepatic function: total bilirubin (TBIL) ≤1.5 times the upper limit of normal value (ULN), or total bilirubin > ULN, but direct bilirubin ≤ULN, ALT, AST ≤2.5 times the upper limit of normal value; Renal function: serum creatinine ≤1.5 times of ULN; Coagulation function: international normalized ratio (INR) or prothrombin time (PT) or activated partial thromboplastin time (aPTT) ≤1.5 x ULN;
* 6. The electrocardiograph was generally normal, and the left ventricular ejection fraction (LVEF) was ≥50%, Or the myocardial enzyme spectrum is in the normal range;
* 7. Normal thyroid function, defined as thyroid-stimulating hormone (TSH) in the normal range; If baseline TSH is beyond the normal range, subjects with total T3 (or FT3) and FT4 in the normal range will also be enrolled;
* 8. Female subjects of childbearing potential have a negative pregnancy test and must agree to take effective contraceptive measures during the study period and within 3 months after the last dose;
* 9. Be willing and able to provide written informed consent/assent for the trial.

Exclusion Criteria:

* 1. Patients with possible tracheoesophageal fistula or aortic esophageal fistula;
* 2. Patients with active autoimmune disease or documented autoimmune disease or symptoms requiring systemic hormone therapy or anti-autoimmune drug therapy;
* 3. Patients with immunodeficiency or who were still receiving systemic steroid hormone therapy (prednisone > 10 mg/ day or other equivalent drugs) or other forms of immunosuppressive therapy 7 days prior to the first dose of neoadjuvant therapy in this study;
* 4. Received anti-tumor therapy, including but not limited to chemotherapy, radiotherapy, immunotherapy, and targeted therapy, within 28 days prior to initial administration;
* 5. Patients with active infection who still required systemic treatment 7 days before the first dose of neoadjuvant therapy in this study;
* 6. Uncontrolled brain metastases;
* 7. Patients with interstitial lung disease, non-infectious pneumonia, or pulmonary fibrosis;
* 8. Patients with active tuberculosis (TB), who is receiving anti-TB treatment or who has received anti-TB treatment within 1 year before the first drug use
* 9. Patients with uncontrolled diabetes (fasting blood glucose ≥CTCAE level 2);
* 10. Peripheral neuropathy of degree II or above was found within 4 weeks before enrollment;
* 11.Patients who have received a foreign organ or stem cell transplant in the past;
* 12. Patients with allergies to the drugs or related ingredients in this study;
* 13. Patients with any serious or unstable medical condition or mental illness;
* 14. History of drug abuse or dependence;
* 15. Major organ disorders or diseases: liver and kidney dysfunction, history of myocardial infarction, unstable heart disease, chronic active hepatitis, etc;
* 16. History of other malignancies within 5 years (except for cured cervical cancer or basal cell carcinoma of the skin);
* 17. Patients who also participated in other clinical trials;
* 18. The researchers did not consider the patients suitable for any medical condition under study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with esophageal squamous cell carcinoma who accept esophagectomy alone or neoadjuvant chemoradiotherapy treatment followed by surgery are acceptable.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete pathologic response rate and its relationship between peripheral blood of lymphocyte and immunocyte. | 3 months
  Definition of complete pathologic response is "no cancer cell, including lympho nodes".
Postoperative pulmonary infection rate and its relationship between peripheral blood of lymphocyte and immunocyte. | 3 months
  The pulmonary infection after surgery included bacterial pneumonia and viral pneumonia and fungal pneumonia.

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Cancer Hospital and Research Institute, Chengdu, Sichuan, China